CLINICAL TRIAL: NCT02896556
Title: Evaluation of Esthetic Performance of Resin Infiltration Technique on Hypomineralized and Demineralized Enamel Lesions
Brief Title: Evaluation of Esthetic Performance of Resin Infiltration Technique on Enamel Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUDHF-2-Icon
Record Dates: First submitted 2016-08-25; First posted 2016-09-12 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Tooth Demineralization
Keywords: image analysis
MeSH Terms: conditions — Tooth Demineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resin infiltrate (Experimental): This is a single-arm study. Resin infiltration technique will be performed to all patients.
  Interventions: Device: Resin infiltrate

INTERVENTIONS:
Device: Resin infiltrate — A resin that used for micro-invasive treatment of enamel-restricted, non-cavitated caries or hypo/demineralized smooth enamel surfaces.

SUMMARY:
The purpose of this study is to evaluate the esthetic performance of resin infiltration technique on superficial hypo-mineralized and demineralized enamel lesions of anterior teeth

DETAILED DESCRIPTION:
The teeth that meet the inclusion criteria will be cleaned from debris and clinical intra-oral photos of the lesions will be taken before and after the treatment. Resin infiltration technique will be performed according to manufacturer's instructions under rubber-dam isolation. Intra-oral photos will be taken directly after infiltration (1 day), and 1 week and 6 months later.

The system of the Commission Internationale de l'Eclairage (CIE) involving 3 color parameters: lightness (L), red/ green chromaticity (a), and yellow/blue chromaticity (b), will be used to assess the extent and durability of color and lightness changes between lesion and sound enamel areas before and after resin infiltration. The extent of assimilation and durability of effect will be assessed by comparing CIE L*a*b data collected before infiltration (baseline), directly after infiltration (1 day), and 1 week and 6 months later.

The color assessments were standardized using a spectrophotometer (SpectroShade, Italy). Lesion areas will be measured for each time point by using an image analysis toolkit (ImageJ, National Institutes of Health, Bethesda, Md.).

Multifactorial analysis of variance with repeated measures will be used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parents of patients who accept to participate and sign the informed consent.
* At least one non-cavitated anterior teeth with a superficial discoloration on enamel due to demineralization or hypo mineralization
* Fully erupted anterior teeth with closed apices.

Exclusion Criteria:

* Patients and parents of patients who accept to participate.
* Teeth having absence of active cavitated-caries lesions, root canal treatment or restorations
* Teeth with ICDAS code 3 lesions (localized enamel breakdown due to caries with no visible dentin)
* Teeth that have a previously esthetic procedure (e.g. bleaching)
* Patients who are not in cooperation with the procedure.
* Fully erupted teeth with open apices

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Esthetic success of resin-infiltration technique after 6 months as assessed by spectrophotometry | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zafer C Cehreli, Prof, Principal Investigator — zcehreli@gmail.com
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim S, Kim EY, Jeong TS, Kim JW. The evaluation of resin infiltration for masking labial enamel white spot lesions. Int J Paediatr Dent. 2011 Jul;21(4):241-8. doi: 10.1111/j.1365-263X.2011.01126.x. Epub 2011 Mar 14. PMID 21401750
- [Background] Knosel M, Eckstein A, Helms HJ. Durability of esthetic improvement following Icon resin infiltration of multibracket-induced white spot lesions compared with no therapy over 6 months: a single-center, split-mouth, randomized clinical trial. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):86-96. doi: 10.1016/j.ajodo.2013.02.029. PMID 23810050
- [Background] Senestraro SV, Crowe JJ, Wang M, Vo A, Huang G, Ferracane J, Covell DA Jr. Minimally invasive resin infiltration of arrested white-spot lesions: a randomized clinical trial. J Am Dent Assoc. 2013 Sep;144(9):997-1005. doi: 10.14219/jada.archive.2013.0225. PMID 23989837